CLINICAL TRIAL: NCT02375542
Title: Clinical Observation and Pathological Characterization of Aortic Tissue at Reoperation
Brief Title: Characterization of Aortic Tissue at Reoperation
Status: Completed | Type: Observational
Sponsor: CryoLife Europa (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO1301.001M
Record Dates: First submitted 2014-08-19; First posted 2015-03-02 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Aortic Aneurysm; Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of aortic tissue which are removed as standard practice during surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Reoperation: Patients who have previously undergone a cardiac operation with the use of BioGlue and are now undergoing a reoperation

SUMMARY:
This study will analyse factors contributing to cardiac re-operation to determine causative effects

DETAILED DESCRIPTION:
This study will collect clinical data on the characteristics of aortic tissue on which BioGlue has been applied during a previous cardiovascular surgery. This is a post market surveillance study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing an aortic re-operation
* Subject has had BioGlue used during previous aortic surgery
* Subject is willing and able to give written informed consent for participation

Exclusion Criteria:

* Subject with a history of vasculitis
* Subject with active infection (endocarditis)
* Subject with a history of chronic inflammatory condition which may have led to ongoing tissue damage
* Subject with a history of auto immune disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective, Single center, single arm study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The microscopic evaluation of the presence of BioGlue on aortic tissue | "participants will be followed for the duration of their surgery, an expected average of 5 hours

SECONDARY OUTCOMES:
Observation and characterization of BioGlue usage during the reoperation procedure | "participants will be followed for the duration of their surgery, an expected average of 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Davide Pacini, Dr, Principal Investigator — Cardiac Surgeon
Locations (1):
- S.Orsola Malpighi Hospital, Bologna, Italy